CLINICAL TRIAL: NCT01631448
Title: Application of the Biological Fibrin Based Adhesive for the Prevention of Surgical Complications in the Kidney Transplant
Brief Title: Fibrin Based Adhesive for the Prevention of Surgical Complications in the Kidney Transplantation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alejandro Gonzalez-Ojeda (Other Government)
Responsible Party: Sponsor-Investigator, Alejandro Gonzalez-Ojeda, PhD, Instituto Mexicano del Seguro Social
Organization: Instituto Mexicano del Seguro Social (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Fibrin-2012-01
Record Dates: First submitted 2012-06-27; First posted 2012-06-29 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2015-03

CONDITIONS: Vascular Postoperative Complications; Urological System Complication of Procedure; Lymphocele; Postoperative Infection
Keywords: Fibrin sealant; renal transplantation; surgical complication
MeSH Terms: conditions — Lymphocele | interventions — Fibrin Tissue Adhesive

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): Patients fron this group do not receive the fibrin sealant
- Fibrin group (Active Comparator): Patients from this group will receive the fibrin sealant
  Interventions: Biological: Fibrin Glue

INTERVENTIONS:
Biological: Fibrin Glue — The biological adhesive will be applied to the study group, with the spray technique in two atmospheres of pressure in a total amount of 10 ml.
  Other Names: Tissucol 10 ml (Baxter)
  Arms: Fibrin group

SUMMARY:
Globally there have been about 45,000 kidney transplants last year. Currently, the overall survival of renal transplant receptors is 95% in the first year and 85% at 5 years. A major challenge to overcome by the renal transplant surgeons, are surgical complications which may impact on patient morbidity and mortality, as well as graft function.

The aim of the study is to assess whether application of fibrin seal prevents postoperative complications in patients undergoing kidney transplantation.

Controlled clinical trial with single-blind evaluation in patients surgically intervened kidney transplantation. It will include all patients undergoing renal transplantation in this Medical Center, any gender and over than 16 years and under 60 years.

DETAILED DESCRIPTION:
INTRODUCTION:

Globally there have been about 45,000 kidney transplants last year. Currently, the overall survival of renal transplant receptors is 95% in the first year and 85% at 5 years. A major challenge to overcome by the renal transplant surgeons, are surgical complications which may impact on patient morbidity and mortality, as well as graft function.

Since 2000 to date the specialties Hospital from the Western Medical Center of the Mexican Institute of Social Security, is the hospital where the greatest number of kidney transplants are performed, reporting to December 2005 a total of 990 cases, with an average of 200 transplants annually.

Since the completion of the first kidney transplants, there has emerged the presence of complications related to the surgical procedure, which have influenced the morbidity and mortality in transplant patients. Several factors are attributed to the occurrence of postoperative complications, such as the patient's nutritional status, ischemic time, presence of comorbidities, organ preservation, surgical technique, experience and skills of the surgeon and the postoperative care.

The main causes of complications in the kidney transplants are: urological complications such as urinary fistula, ureteral obstruction and ureteral necrosis (less than 7% of all kidney transplants). Ischemia is the most common probable cause of urological complications secondary to donor kidney extraction, anastomotic technique, variations in vascular supply, rejection or medication. Vascular complications as early arterial thrombosis, renal vein thrombosis and renal artery stenosis, are almost always due to a technical complication, or are accompanied by twisting or bending of blood vessels during placement of the transplanted kidney. Technical difficulties may be secondary to atherosclerotic disease in the donor or receptor, or interact with multiple arteries. Lymphatic complications as lymphocele and lymphatic fistula, after renal transplantation accumulation of lymphatic fluid postoperatively are up to 15% of the patients. It is believed that the origin of the lymph is in the destruction of perivascular normal lymph ducts during dissection, or destruction of the hilar lymph.

Decreasing the incidence of surgical wound infection after renal transplantation is multifactorial and is related to advances in the treatment of anemia, uremia, and general health of patients with end-stage renal disease.

The seals are partly fibrin blood products and pharmacological agents. Their specific use is as an adjunct to hemostasis as tissue adhesive. Seals are also developed as fibrin vehicle to provide antimicrobial pharmacological agents, chemotherapeutic agents and growth factors.

They have the advantage of being products of human origin without tissue toxicity, which promotes rapid fibrin seal. The seal is normally reabsorbed in days, promoting local tissue growth and repair without increasing perioperative development of adhesions.

OBJECTIVE:

Assess whether application of fibrin seal prevents postoperative complications in patients undergoing kidney transplantation.

MATERIAL AND METHODS:

Controlled clinical trial with single-blind evaluation in patients surgically intervened kidney transplantation. It will include all patients undergoing renal transplantation in this Medical Center, any gender and over than 16 years and under 60 years. Patients will be excluded with allergy to the fibrin glue components. All the transplant procedure will be made for the same surgical team.

The receptor site preparation will be done by addressing the retroperitoneal region of the right lower quadrant of the abdomen with an incision Gibson type.

The patients are going to be distributed into two groups: Group 1: fibrin, Group 2: Control. Complication weather vascular, urological, lymphatic, infectious, hospital stay and graft loss will be assessed.

The receptor site preparation will be done by addressing the retroperitoneal region of the right lower quadrant of the abdomen with an incision Gibson type.

The dissection of great vessels will be performed to achieve hemostasis of the blood vessels and nodes, with electrocoagulation and ligation gauge nonabsorbable 3-0.

The vascular anastomosis will be made to the external iliac vessels of the receptor in shaped end-side way, the suture material in size 6-0, in continuous sutures type with nonabsorbable monofilament. The new ureteral anastomosis will be performed with the modified technique of Leriche-Gregoire.

The new ureter will be tunneled and anastomosed to the mucosa with absorbable suture material 4-0 (polyglactin). The biological adhesive will be applied to the study group, with the spray technique in two atmospheres of pressure in a total amount of 10 ml. No biological adhesive, placebo or simulated technique will be performed to the control group.

There will be placed a continuous suction drainage of closed silicone type, and the abdominal wall will be closed with absorbable material in both groups.

Patients will be followed from the immediate postoperative period until discharge, and at follow up every week the first month, then every 15 days the second month, and monthly until one year follow up. During this follow-up, patients will be assessed through laboratory tests that include complete blood count, blood chemistry with serial measurements of serum creatinine, glomerular filtration rate, serum electrolytes and blood levels of immunosuppressants. Also patients will be followed from the clinical point of view and if there is any suspect for a complication, laboratory exams will be conducted such as crops, urinalysis, determination of creatinine, noninvasive imaging studies such as Doppler ultrasound, computed tomography, angiography if suspect on vascular complications.

STATISTICAL ANALYSIS:

Nominal variables were analyzed using percentage frequencies, X2 test or Fisher exact test. Numeric variables using Student's t test for independent samples and ANOVA with post hoc Scheffe test. U Mann Whitney and Kruskal Wallis tests will be used as long as data do not conform to normal distribution.

ELIGIBILITY:
Inclusion Criteria:

* Patients candidates to renal transplantation

Exclusion Criteria:

* Patients with known allergy to products of fibrin seal

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 152 (Actual)
Dates: Start 2010-05; Primary Completion 2014-01 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Postoperative Complications | 1 year
  Patients will be followed from the immediate postoperative period until discharge, and at follow up every week the first month, then every 15 days the second month, and monthly until one year follow up. Identifying any kind of complication derived from the surgical procedure.

SECONDARY OUTCOMES:
Vascular Postoperative Complications | 1 year
  Identifying the different possible vascular postoperative complications:
  * Renal artery stenosis: The narrowing of the light by 30% diagnosed by Doppler ecosonography and corroborated by arteriography.
  * Renal vein stenosis: The narrowing of light> 40% of the renal vein Doppler and confirmed by venography ecosonography graft.
  * Arterial thrombosis: The total occlusion of the renal artery lumen by a thrombus, which prevents blood perfusion of the kidney, diagnosed by Doppler and arteriography of the graft.
Urological System Complication of Procedure | 1 year
  Identifying the different possible urological postoperative complications:
  * Urinary Fistula: The loss of continuity of the ureterovesical anastomosis with formation of a journey outward, allowing the escape of urine into the preperitoneal region at the site of graft placement.
  * Ureteral obstruction: Stopping or reducing the passage of urine into the bladder through the ureter at the ureterovesical anastomosis, which is given by hyperplasia at the site.
  * Ureteral necrosis: devitalization of the ureter as a result of devascularization, with loss of functionality and feasibility.
Lymphocele | 1 year
  Identifying the different possible lymphatic postoperative complications:
  * Lymphocele: encapsulated collection of lymphatic fluid in postoperative graft site.
  * Lymphatic fistula: Leakage of lymph fluid with formation of a journey to the outside of the surgical wound.
Postoperative Infection | 1 year
  Identifying the different possible infectious postoperative complications:
  *Surgical wound infection: Signs of wound infection, like redness, heat, increased local temperature and swelling of the wound. If the drain or treat this is limited, the subcutaneous tissue infection was considered superficial infection of the surgical site, if any collection of pus in the thickness of wound without involvement of the surgical wound abscess be known. If there is necrosis necrotizing myofasciitis be called.

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro Gonzalez-Ojeda, PhD, Study Director — Instituto Mexicano del Seguro Social
Locations (2):
- Mexico (2):
  - Department of Transplantation. Specialties Hospital. Mexican Institute of Sociaql Security, Guadalajara, Jalisco
  - Research Unit in Clinical Epidemiology, Specialties Hospital. Mexican Institute of Social Security, Guadalajara, Jalisco